CLINICAL TRIAL: NCT01411319
Title: A Phase I Trial of MRI-Guided Lattice Extreme Ablative Dose Radiotherapy For Prostate Cancer
Brief Title: MRI-Guided Lattice Extreme Ablative Dose Radiotherapy For Prostate Cancer
Acronym: LEAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alan Pollack, MD, PhD, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20100389; R21CA153826 (NIH)
Record Dates: First submitted 2011-08-03; First posted 2011-08-08 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- LEAD Radiation Therapy (Experimental): Participants in this group will receive the LEAD Radiation Therapy on Day 1 followed by 38 daily standard IMRT beginning Day 2.
  Interventions: Radiation: Lattice Extreme Ablative Dose Radiation Therapy; Radiation: Standard IMRT

INTERVENTIONS:
Radiation: Lattice Extreme Ablative Dose Radiation Therapy — 12 - 14 Gy dose pipes in 1 fraction to the multiparametric MRI defined gross tumor volumes (GTV) on Day 1.
  Other Names: LEAD RT
Radiation: Standard IMRT — 76 Gy in 38 fractions (2 Gy daily) of Standard Intensity-modulated radiation therapy (IMRT) starting on Day 2 for 7.5 weeks.
  Other Names: IMRT

SUMMARY:
The hypotheses of this study are:

1. Delivery of single fraction Lattice Extreme Ablative Dose (LEAD) radiotherapy (RT) to the dominant tumor lesion(s) in the prostate as identified by multiparametric functional Magnetic Resonance Imaging is safe and feasible when given prior to standard prostate radiotherapy.
2. Biomarker expression levels differ in the functional MRI identified suspicious tumor regions and unsuspicious tumor regions. The investigators hypothesize that a significant source of variation in biomarker levels is due to tumor heterogeneity and that it is molecular abnormalities in the dominant tumor areas that are angiogenic and determine outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy confirmed adenocarcinoma of the prostate.
2. T1-T3a disease based on digital rectal exam (DRE).

   * T3a disease based on MRI is acceptable (no evidence of frank (clear cut) seminal vesicle (SV) involvement or invasion of bladder or rectum).
3. Gleason score 6-10.
4. Patients with Gleason score ≥8 must be offered long term androgen deprivation therapy (ADT) and refuse such treatment because only 4-6 months (+/- 2 months) (short term ADT) is permitted (not required) on this protocol. The ADT is recommended to begin after fiducial marker placement; however, ADT is permitted to have been started up to two months prior to the signing of consent. All patients in this protocol may (not required) be treated with 4-6 months (+/- 2 months) of ADT, at the discretion of the treating physician.

   * Gleason ≥ 8 must have < 40% of the tissue involved with Gleason 8 in the biopsy specimen.
5. Prostate-specific antigen (PSA) ≤ 30 ng/mL within 3 months of enrollment. If PSA was above 30 and dropped to ≤ 30 with antibiotics, this is acceptable for enrollment.
6. No previous pelvic radiotherapy.
7. No previous history of radical/total prostatectomy (suprapubic prostatectomy is acceptable).
8. No concurrent, active malignancy, other than nonmetastatic skin cancer or early stage chronic lymphocytic leukemia (well-differentiated small cell lymphocytic lymphoma). If a prior malignancy is in remission for ≥ 5 years then the patient is eligible.
9. Identifiable multiparametric-MRI tumor lesion or lesions, that total in volume < 33% of the prostate

   * Multiparametric MRI of prostate and pelvis is required prior to protocol consideration.
   * If contrast not given, the point dose on the apparent diffusion coefficient (ADC) map should be < 1000.
10. Ability to understand and the willingness to sign a written informed consent document.
11. Zubrod performance status < 2.
12. Willingness to fill out quality of life forms.
13. Bone scan negative if PSA > 15 ng/mL or Gleason ≥ 8 disease. A questionable bone scan is acceptable if other imaging tests are negative for metastasis.
14. Serum testosterone is within 40% of normal assay limits (e.g., x=0.4*lower assay limit and x=.04*upper assay limit + upper assay limit), and taken within 4 months of enrollment. Patients who have been started on ADT prior to signing consent are not required to have a serum testosterone at this level prior to signing consent; but, a serum testosterone prior to fiducial marker placement is recommended.
15. Serum liver function tests (LFT) are taken within 3 months of enrollment.
16. Complete blood counts are taken within 3 months of enrollment.
17. Age ≥ 35 and ≤ 85 years.

Exclusion Criteria:

1. > T3a disease on digital rectal exam or >T3a disease clearly identified by MRI.
2. Gleason score < 6.
3. ≥ 40% Gleason 8-10 tumor, over the total tissue including other tumor and normal tissue. For example: (Gleason 8-10 tumor length/other biopsy tissue length)*100 = ≥ 40%.
4. Androgen deprivation therapy longer than 8 months. Androgen deprivation timing is for the Luteinizing hormone-releasing hormone (LHRH) agonist portion only and not when anti-androgen is started beforehand with the purpose of counteracting the surge in testosterone from the LHRH agonist - PSA > 30 ng/mL within 3 months of enrollment.
5. PSA > 30 ng/mL within 3 months of enrollment
6. Unable to obtain a 1.5T or 3.0T multiparametric MRI of the pelvis and prostate with contrast.
7. Unidentifiable multiparametric MRI tumor lesion.
8. Identifiable multiparametric-MRI tumor lesions, that total in volume ≥ 33% of the prostate.
9. Previous pelvic radiotherapy.
10. Previous history of radical prostatectomy.
11. Concurrent, active malignancy, which is not nonmetastatic skin cancer or early stage chronic lymphocytic leukemia (well-differentiated small cell lymphocytic lymphoma). If a prior malignancy is in remission for < 5 years then the patient is not eligible.
12. Zubrod performance status ≥ 2.
13. Inability to understand or unwilling to sign a written informed consent document
14. Unwilling to fill out quality of life/psychosocial forms.
15. Bone scan is positive and other imaging tests confirm a suspicion of metastasis from prostate cancer.
16. Serum testosterone is not within 40% of normal assay limits taken within 4 months of enrollment (only applicable to patients not started on ADT prior to signing consent).
17. Serum liver function tests (LFTs) are not taken within 3 months of enrollment.
18. Complete blood counts are not taken within 3 months of enrollment.
19. Age < 35 and > 85 years.

Ages: 35 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-12-27 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2020-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Pollack, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pollack A, Chinea FM, Bossart E, Kwon D, Abramowitz MC, Lynne C, Jorda M, Marples B, Patel VN, Wu X, Reis I, Studenski MT, Casillas J, Stoyanova R. Phase I Trial of MRI-Guided Prostate Cancer Lattice Extreme Ablative Dose (LEAD) Boost Radiation Therapy. Int J Radiat Oncol Biol Phys. 2020 Jun 1;107(2):305-315. doi: 10.1016/j.ijrobp.2020.01.052. Epub 2020 Feb 19. PMID 32084522

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LEAD Radiation Therapy
Started | 25
Completed | 24
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | LEAD Radiation Therapy
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 18
Age, Continuous [Median (Full Range); unit: years] | 67 [44 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Study Participants Experiencing Treatment-Related Toxicity
Description: Toxicity are any Grade 2 or higher treatment-related adverse events as assessed by treating physician using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.0.
Time Frame: Up to 8.5 weeks
Population: All 25 participants were evaluated up to 8.5 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | LEAD Radiation Therapy
Number analyzed (Participants) | 25
Participants
  Serious Adverse Events (SAEs) with Definite Relation to Study Treatment | 0
  SAEs with Probable Relation to Study Treatment | 0
  SAEs with Possible Relation to Study Treatment | 1
  Adverse Events (AEs) with Definite Relation to Study Treatment | 9
  AEs with Probable Relation to Study Treatment | 10
  AEs with Possible Relation to Study Treatment | 5

2. Primary Outcome: Percentage of Enrolled Patients for Whom LEAD RT Dose Can be Successfully Administered Following MRI-guided Planning.
Description: The percentage of enrolled patients for whom LEAD RT dose can be successfully administered following MRI-guided planning.
Time Frame: Up to 8 weeks
Population: All 25 enrolled participants completed the duration of study treatment (8 weeks).
Measure: Number; unit: percentage of participants
Arm/Group | LEAD Radiation Therapy
Number analyzed (Participants) | 25
percentage of participants | 100

3. Secondary Outcome: Number of Participants With Remaining Tumor Cells in the Prostate Post Treatment
Description: The number of participants with positive tumor cells left in the prostate after LEAD RT as evaluated by prostate biopsy.
Time Frame: Up to 2.5 Years
Population: Endpoint biopsy was collected only on 12 of 25 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | LEAD Radiation Therapy
Number analyzed (Participants) | 12
Participants | 1

4. Secondary Outcome: Percentage of Participants With Positive Prostate Biopsies After Completion of Treatment
Description: Preliminary indication of efficacy of treatment will be reported as the percentage of participants with positive prostate biopsies after completion of treatment.
Time Frame: From Baseline to 2.5 Years Post Completion of Study Therapy (Approximately 3 years)
Population: One participant was lost to follow-up at the follow-up period post-completion of treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LEAD Radiation Therapy
Number analyzed (Participants) | 24
percentage of participants | 4 [0.7 to 19.5]

5. Secondary Outcome: Rate of Participants That Achieve Failure-Free Survival (FFS)
Description: The percentage of participants achieving FFS will be reported. Failure-free is defined as no documented evidence of biochemical and/or or clinical failure or death from any cause, whichever occur first. Biochemical failure is defined is a increase of 2 or greater from nadir of Prostate Specific Antigen (PSA) levels. Clinical Failure is defined as newly identified extension outside the prostate after initial regression, or urinary obstructive symptoms with carcinoma or regional/distant failure due to radiographic evidence metastasis.
Time Frame: Up to 6 years
Population: One participant was lost to follow-up at the follow-up period post-completion of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | LEAD Radiation Therapy
Number analyzed (Participants) | 24
percentage of participants | 90.5

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the elapsed time from study enrollment to death from any cause. For surviving patients, follow-up will be censored at the date of last contact.
Time Frame: Up to 6 years
Population: Timeframe allows for study visit windows.
Measure: Median (Full Range); unit: months
Arm/Group | LEAD Radiation Therapy
Number analyzed (Participants) | 25
months | 66 [20.7 to 70.6]

7. Secondary Outcome: HrQoL as Assessed by EPIC-SF12 Questionnaire
Description: Health-related Quality of Life (HRQOL) will be measured using the Expanded Prostate Cancer Index Composite and Medical Outcomes Study SF-12 (EPIC SF-12) to evaluate patient function and satisfaction after prostate cancer treatment. The questionnaire has 5 subscales (Urinary Function, Urinary Symptoms, Bowel Habits, Sexual Function and Hormonal Function). Each subscale has a total score ranging from 0-100, with higher scores representing better HRQOL.
Time Frame: At Baseline (Prior to RT), at 8 weeks (Last week of RT), At 6 weeks post RT, At 3 months post RT, At 6 months post RT, At 9 months post RT, At 15 months post RT, At 27 months post RT, At 39 months post RT, At 51 months post RT, At 63 months post RT
Population: Not all participants were able to complete the questionnaires at different timepoints in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LEAD Radiation Therapy
Number analyzed (Participants) | 25
score on a scale
  Urinary Function: Prior to Radiation Therapy (RT) | 94.5 (10.9)
  Urinary Function: 8 Weeks (Last Week of RT) | 92.5 (14.4)
  Urinary Function: 6 Weeks Post-RT: number analyzed (Participants) | 24
  Urinary Function: 6 Weeks Post-RT | 92.8 (20)
  Urinary Function: 3 Months Post-RT: number analyzed (Participants) | 23
  Urinary Function: 3 Months Post-RT | 93.1 (17.6)
  Urinary Function: 9 Months Post-RT: number analyzed (Participants) | 22
  Urinary Function: 9 Months Post-RT | 93.5 (16.6)
  Urinary Function: 15 Months Post-RT: number analyzed (Participants) | 22
  Urinary Function: 15 Months Post-RT | 93.2 (14.5)
  Urinary Function: 27 Months Post-RT: number analyzed (Participants) | 20
  Urinary Function: 27 Months Post-RT | 93.6 (15.5)
  Urinary Function: 39 Months Post-RT: number analyzed (Participants) | 18
  Urinary Function: 39 Months Post-RT | 95.8 (9.2)
  Urinary Function: 51 Months Post-RT: number analyzed (Participants) | 17
  Urinary Function: 51 Months Post-RT | 92.8 (17)
  Urinary Function: 63 Months Post-RT: number analyzed (Participants) | 17
  Urinary Function: 63 Months Post-RT | 94.2 (18.8)
  Urinary Symptoms: Prior to RT | 88.5 (13.9)
  Urinary Symptoms: 8 Weeks (Last Week of RT): number analyzed (Participants) | 24
  Urinary Symptoms: 8 Weeks (Last Week of RT) | 79.2 (13)
  Urinary Symptoms: 6 Weeks Post-RT: number analyzed (Participants) | 24
  Urinary Symptoms: 6 Weeks Post-RT | 85.7 (11.9)
  Urinary Symptoms: 3 Months Post-RT: number analyzed (Participants) | 23
  Urinary Symptoms: 3 Months Post-RT | 87.5 (11.6)
  Urinary Symptoms: 9 Months Post-RT: number analyzed (Participants) | 21
  Urinary Symptoms: 9 Months Post-RT | 85.1 (17.9)
  Urinary Symptoms: 15 Months Post-RT: number analyzed (Participants) | 23
  Urinary Symptoms: 15 Months Post-RT | 87.2 (13.8)
  Urinary Symptoms: 27 Months Post-RT: number analyzed (Participants) | 19
  Urinary Symptoms: 27 Months Post-RT | 91.4 (7.3)
  Urinary Symptoms: 39 Months Post-RT: number analyzed (Participants) | 17
  Urinary Symptoms: 39 Months Post-RT | 90.8 (7.4)
  Urinary Symptoms: 51 Months Post-RT: number analyzed (Participants) | 17
  Urinary Symptoms: 51 Months Post-RT | 91.2 (13.6)
  Urinary Symptoms: 63 Months Post-RT: number analyzed (Participants) | 17
  Urinary Symptoms: 63 Months Post-RT | 90.8 (8.6)
  Bowel Habits: Prior to RT | 98.5 (4.5)
  Bowel Habits: 8 Weeks (Last Weeks of RT) | 89.7 (14.1)
  Bowel Habits: 6 Weeks Post-RT: number analyzed (Participants) | 23
  Bowel Habits: 6 Weeks Post-RT | 95.3 (8)
  Bowel Habits: 3 Months Post-RT: number analyzed (Participants) | 23
  Bowel Habits: 3 Months Post-RT | 93.7 (10)
  Bowel Habits: 9 Months Post-RT: number analyzed (Participants) | 22
  Bowel Habits: 9 Months Post-RT | 95.1 (8.3)
  Bowel Habits: 15 Months Post-RT: number analyzed (Participants) | 23
  Bowel Habits: 15 Months Post-RT | 95.7 (6.6)
  Bowel Habits: 27 Months Post-RT: number analyzed (Participants) | 20
  Bowel Habits: 27 Months Post-RT | 93.3 (9.6)
  Bowel Habits: 39 Months Post-RT: number analyzed (Participants) | 18
  Bowel Habits: 39 Months Post-RT | 95.8 (7.6)
  Bowel Habits: 51 Months Post-RT: number analyzed (Participants) | 17
  Bowel Habits: 51 Months Post-RT | 91.7 (13.3)
  Bowel Habits: 63 Months Post-RT: number analyzed (Participants) | 17
  Bowel Habits: 63 Months Post-RT | 93.6 (10.1)
  Sexual Function: Prior to RT: number analyzed (Participants) | 24
  Sexual Function: Prior to RT | 55.2 (23.9)
  Sexual Function: 8 Weeks (Last Week of RT): number analyzed (Participants) | 24
  Sexual Function: 8 Weeks (Last Week of RT) | 39.5 (31.6)
  Sexual Function: 6 Weeks Post-RT: number analyzed (Participants) | 23
  Sexual Function: 6 Weeks Post-RT | 38.2 (34.7)
  Sexual Function: 3 Months Post-RT: number analyzed (Participants) | 20
  Sexual Function: 3 Months Post-RT | 42.7 (37.3)
  Sexual Function: 9 Months Post-RT: number analyzed (Participants) | 22
  Sexual Function: 9 Months Post-RT | 44.6 (33)
  Sexual Function: 15 Months Post-RT: number analyzed (Participants) | 22
  Sexual Function: 15 Months Post-RT | 49.2 (31.4)
  Sexual Function: 27 Months Post-RT: number analyzed (Participants) | 20
  Sexual Function: 27 Months Post-RT | 44.5 (28.8)
  Sexual Function: 39 Months Post-RT: number analyzed (Participants) | 18
  Sexual Function: 39 Months Post-RT | 41.8 (29.2)
  Sexual Function: 51 Months Post-RT: number analyzed (Participants) | 17
  Sexual Function: 51 Months Post-RT | 47.7 (29)
  Sexual Function: 63 Months Post-RT: number analyzed (Participants) | 16
  Sexual Function: 63 Months Post-RT | 36.6 (25.1)
  Hormonal Function: Prior to RT | 88 (15.1)
  Hormonal Function: 8 Weeks (Last week of RT) | 86.2 (15.1)
  Hormonal Function: 6 Weeks Post-RT: number analyzed (Participants) | 24
  Hormonal Function: 6 Weeks Post-RT | 86.5 (13.4)
  Hormonal Function: 3 Months Post-RT: number analyzed (Participants) | 23
  Hormonal Function: 3 Months Post-RT | 85.4 (17.1)
  Hormonal Function: 9 Months Post-RT: number analyzed (Participants) | 22
  Hormonal Function: 9 Months Post-RT | 89.8 (11.4)
  Hormonal Function: 15 Months Post-RT: number analyzed (Participants) | 23
  Hormonal Function: 15 Months Post-RT | 92.8 (9)
  Hormonal Function: 27 Months Post-RT: number analyzed (Participants) | 20
  Hormonal Function: 27 Months Post-RT | 93.8 (7.2)
  Hormonal Function: 39 Months Post-RT: number analyzed (Participants) | 18
  Hormonal Function: 39 Months Post-RT | 91.9 (10.3)
  Hormonal Function: 51 Months Post-RT: number analyzed (Participants) | 17
  Hormonal Function: 51 Months Post-RT | 87.9 (17.1)
  Hormonal Function: 63 Months Post-RT: number analyzed (Participants) | 17
  Hormonal Function: 63 Months Post-RT | 91.5 (10)

8. Secondary Outcome: HrQoL as Assessed by MAX-PC Questionnaire
Description: Health-related quality of life (HRQOL) will be measured using the scores on the Modified 18-item Memorial Anxiety Scale for Prostate Cancer (MAX-PC) from pre-treatment to post-treatment. The scale consists of 18 items (e.g. "I thought about prostate cancer even though I didn't mean to.") scored on a scale from 0 ("not at all") to 3 ("often"). Total scores range from 0 to 54, with higher scores indicating higher levels of anxiety.
Time Frame: as for outcome 7
Population: Not all participants were able to complete the questionnaires at different timepoints in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LEAD Radiation Therapy
Number analyzed (Participants) | 25
score on a scale
  Prior to Radiation Therapy (RT): number analyzed (Participants) | 23
  Prior to Radiation Therapy (RT) | 13.7 (6.3)
  8 Weeks (Last Week of RT) | 15.1 (7.2)
  6 Weeks Post-RT: number analyzed (Participants) | 24
  6 Weeks Post-RT | 13.3 (7.5)
  3 Months Post-RT: number analyzed (Participants) | 22
  3 Months Post-RT | 11.7 (7.5)
  9 Months Post-RT: number analyzed (Participants) | 22
  9 Months Post-RT | 12.6 (7.5)
  15 Months Post-RT: number analyzed (Participants) | 23
  15 Months Post-RT | 10 (6.9)
  27 Months Post-RT: number analyzed (Participants) | 20
  27 Months Post-RT | 12.2 (6.1)
  39 Months Post-RT: number analyzed (Participants) | 18
  39 Months Post-RT | 12.3 (7.2)
  51 Months Post-RT: number analyzed (Participants) | 17
  51 Months Post-RT | 11.2 (9.1)
  63 Months Post-RT: number analyzed (Participants) | 17
  63 Months Post-RT | 12.9 (6.2)

ADVERSE EVENTS:
Time Frame: Up to 6 years
Arm/Group | LEAD Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEAD Radiation Therapy (N=25)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEAD Radiation Therapy (N=25)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
Low Testosterone (Blood and lymphatic system disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4)
Cystitis noninfective (Renal and urinary disorders) | 13 (17)
Diarrhea (Gastrointestinal disorders) | 9 (15)
Dizziness (Nervous system disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Ejaculation disorder (Reproductive system and breast disorders) | 1 (1)
Low Testosterone (Endocrine disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 3 (5)
Fatigue (General disorders) | 10 (11)
Fever (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Increased appetite (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 3 (3)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Low testosterone (Investigations) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Prostatic pain (Reproductive system and breast disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 4 (4)
Urinary obstructive symptoms, urinary hesitancy, increased frequency of bowel movement (no diarrhea) (Renal and urinary disorders) | 7 (7)
Urinary frequency (Renal and urinary disorders) | 19 (27)
Urinary incontinence (Renal and urinary disorders) | 4 (4)
Urinary retention (Renal and urinary disorders) | 8 (9)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 4 (5)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 16 (25)
Weight loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT01411319/Prot_SAP_000.pdf